CLINICAL TRIAL: NCT00748072
Title: 1-deamino 8-d-arginine Vasopressin in Percutaneous Ultrasound-guided Renal Biopsy: a Randomized Controlled Trial
Brief Title: 1-deamino 8-d-arginine Vasopressin (DDAVP) in Percutaneous Ultrasound-guided Renal Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Carlo Manno, Assistant Professor, Chair of Nephrology, Unit of Nephrology, University of Bari, Bari, Italy, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DDAVP 01
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Failure
Keywords: Vasopressin; bleeding; biopsy; ultrasonography
MeSH Terms: conditions — Renal Insufficiency; Diabetes Insipidus; Hemorrhage | interventions — Deamino Arginine Vasopressin; Vasopressins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline solution (Placebo Comparator): patients treated with 1 ml of s.c. saline solution
  Interventions: Drug: saline solution
- DDAVP (Experimental): treated with DDAVP (0.3 mcg/Kg s.c.) 1 hour before renal biopsy
  Interventions: Drug: DDAVP

INTERVENTIONS:
Drug: DDAVP — 0.3 mcg/kg subcutaneous
  Other Names: vasopressin
  Arms: DDAVP
Drug: saline solution — saline solution 1 ml subcutaneous
  Other Names: placebo
  Arms: Saline solution

SUMMARY:
The investigators evaluated the effect of pre-biopsy treatment with 1-deamino-8-D-arginine (DDAVP) on the incidence of post-biopsy bleeding complications. This is a IV phase single centre, double blind, randomized controlled study in patients, with acute and chronic nephropathy, undergoing ultrasound-guided percutaneous renal biopsy.

DETAILED DESCRIPTION:
Renal biopsy is an essential procedure in the diagnosis of primary and secondary renal diseases. The technique has significantly improved over the past two decades because of the introduction of ultrasonography and automated-gun biopsy devices; however an accurate clinical, chemistry and renal ultrasound evaluation before and 24-hours post renal biopsy is necessary, because bleeding complications still occur in about 1/3 of our procedures, with major complications occurring in only 1.2% of patients. Of the data routinely collected for potential predictors of post-biopsy bleeding complications, only gender, age, and baseline partial thromboplastin time show a significant predictive value. The other variables investigated do not have any predictive value (Manno C et al, Kidney Int 2004). The majority of published studies, retrospective and non-randomized, on this topic have focused on the comparative performance of different renal biopsy techniques and types of needles, but no study has shown potential predictors of post-biopsy bleeding complications. On the other hand, the available studies have not shown any specific test to select patients with major risk of post-biopsy bleeding.

The aim of this study is to evaluate the effect of pre-biopsy treatment with DDAVP or desmopressin on the incidence of post-biopsy bleeding complications.

DDAVP is a synthetic derivative of the anti-diuretic hormone vasopressin; therefore, the administration of DDAVP is often accompanied by water retention, a drop in blood pressure and a secondary increase in heart rate. The haemostatic effect of DDAVP is related to an increase of vWF-factor VIII levels. DDAVP is the treatment of choice for most patients with von Willebrand (type I) disease and haemophilia A; moreover, the compound has been shown to be useful in a variety of inherited and acquired hemorrhagic conditions, including some congenital platelet function defects, chronic liver disease, uremia, and haemostatic defects induced by the therapeutic use of anti-thrombotic drugs such as aspirin and ticlopidine. Finally, DDAVP has been used as a haemostatic agent in patients undergoing surgery at major risk of bleeding. Disadvantages of DDAVP include reported rare thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females > 16 and < 80 years of age.
2. Blood pressure < 140/90 mmHg.
3. Serum creatinine ≤ 1.5 mg/dl and/or creatinine clearance ≥ 60 ml/min.
4. Bleeding time, prothrombin time, partial thromboplastin time, platelets and fibrinogen in the normal range.

Exclusion Criteria:

1. Biopsy of transplant kidney
2. Poorly controlled hypertension
3. Single kidney
4. Renal cancer
5. Hydro/pyonephrosis
6. Renal size significantly reduced
7. Severe obesity
8. Coagulation disorder
9. Serum creatinine > 1.5 mg/dl and/or creatinine clearance < 60 ml/min

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Manno, MD, Principal Investigator — University of Bari
Locations (1):
- Center and Atelier for Epidemiological Studies, University of Bari, Bari, Bari, Italy

REFERENCES:
- [Derived] Manno C, Bonifati C, Torres DD, Campobasso N, Schena FP. Desmopressin acetate in percutaneous ultrasound-guided kidney biopsy: a randomized controlled trial. Am J Kidney Dis. 2011 Jun;57(6):850-5. doi: 10.1053/j.ajkd.2010.12.019. Epub 2011 Feb 26. PMID 21354681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled all patients with serum creatinine less than 1.5 mg/dL and/or estimated glomerular filtration rate greater than 60 mL/min/1.73m2 and normal coagulation parameters, undergoing ultrasound-guided biopsy of native kidney, in our Unit, from August 2008 to December 2009.
Pre-assignment Details: The exclusion criteria were solitary kidney, kidney cancer, hydro/pyonephrosis, significantly reduced renal size at ultrasound image, severe obesity (body mass index > 30), chronic kidney disease and acute kidney injury.
Period: Overall Study
Arm/Group | Saline Solution | DDAVP
Started | 82 | 80
Completed | 82 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Solution | DDAVP | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (15.0) | 39.5 (14.2) | 40.6 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was the Incidence of Post-biopsy Bleeding Complications.
Time Frame: Immediately post-biopsy and 24 hours post-biopsy.
Measure: Number; unit: participants
Arm/Group | Saline Solution | DDAVP
Number analyzed (Participants) | 82 | 80
participants | 25 | 11
Statistical Analysis 1: Comparison: Saline Solution vs DDAVP; The sample size was calculated by the difference in post-biopsy bleeding complications. Since the presence of bleeding was demonstrated in about 30-40 % in our previous observational study, we hypothesized a reduction risk of 0.50 and an absolute reduction of risk from 0.40 to 0.20. The sample size of the study for a power of 0.80 and a significance level <0.05 was calculated in 158 patients; Test type: Superiority or Other; p = 0.01, Chi-squared; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.24 to 0.85]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: heart rate was monitored every 6 hours after the biopsy for 24 hours
Arm/Group | Saline Solution | DDAVP
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/80
Other Adverse Events (participants affected / at risk) | 0/82 | 3/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Solution (N=82) | DDAVP (N=80)
mild increase of heart rate (Cardiac disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
A possible limitation of the study is the single-center design of the study, which could reduce the generalizability of our results and their external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes